CLINICAL TRIAL: NCT04073199
Title: Effectiveness of the Stretching of the Teres Major in Patients Suffering From Subacromial Syndrome
Brief Title: Comparison of Two Stretching Techniques in Patients Suffering From Subacromial Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: P17/072
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Subacromial Impingement Syndrome
Keywords: stretching,teres major, subacromial syndrome, manual therapy
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Long Lever Group (Active Comparator): This arm receive the protocolized treatment along with the long passive stretch of the Teres Major in Long Lever with the patient in supine position.
  Interventions: Procedure: Long Lever Group
- Short Lever Group (Active Comparator): This arm receive the protocolized treatment along with the short lever stretch according to the Orthopaedic Manual Therapy of the Teres Major.
  Interventions: Procedure: Short Lever Group
- Control Group (No Intervention): only receive the protocolized physiotherapy treatment for the Subacromial syndrome that is applied in the Rehabilitation Service, without the addition of any additional stretch technique.

INTERVENTIONS:
Procedure: Long Lever Group — the physiotherapist wears the limb passively towards flexion, external rotation and abduction until the physiotherapist has perception of stretch of the tissues (sensation terminal elastic firm according to the concept of Orthopaedic Manual Therapy for the soft tissue treatment) The patient's own weight stabilizes the proximal segment, in case that the scapula is not stable, the physiotherapist fixes with his free hand the scapula.
  The technique will be performed two days a week, at intervals of 20 seconds of technique and 20 rest periods for ten reps (estimated time per session is 7 minutes approximate).
  Arms: Long Lever Group
Procedure: Short Lever Group — It consists of a stretch made by the physiotherapist, with the patient in supine position, with the extremity to be treated in a submaximal position of flexion and external rotation (fixed by the arm and body of the physiotherapist) and realizing the stretch a through the scapula in the medial and caudal dorsal direction.
  The technique will be performed two days per week, at intervals of 20 seconds of technique and 20 rest periods for ten reps (estimated time per session is 7 minutes approximate)
  Arms: Short Lever Group

SUMMARY:
The shoulder stability has always been related to the rotator cuff complex, although more and more is contemplated the Teres Major muscle and its affectation in the shape of the trigger points within this pathology. As non-invasive measures for the deactivation of these myofascial points, Travell and Simons recommended the pressure maintained along with muscular stretch.

Stretching are usually a technique widely used in our practice as physiotherapists and it is necessary to study its effects in the clinic. As an objective we plan to compare the effect of passive stretching in short lever according to the Orthopaedic Manual Therapy concept if it produces better result in the pain, the rank of movement and in the Function, with the effect of stretching by means of a long lever in affected patients of subacromial syndrome.

This is a randomized controlled study with blind evaluator approved by the Ethical Committee of the Institut d'Investigació en atenció Primaria Jordi Gol.

After checking the inclusion and exclusion criteria, you will be asked, voluntarily, that the patient sign informed consent. The variables will then be valued independent and dependent on the study. It will randomly be assigned to one of the three groups in the study. The 3 groups receive the protocolized treatment for the service they consist of In superficial thermotherapy, an educational talk and kinesitherapy. The intervention groups will receive alternate days, with a total of six sessions, the stretch corresponding to the group to which they have been assigned.

In the case of the Long Lever Group, the intervention consists in a rotary stretch through the humerus as a mobile point. And in the case of the Short Lever Group a stretch of translocation through the scapula as a mobile point.

The main variables used will be: age, side effects, habits involving the shoulder, pain intensity, pain threshold at pressure and function, among others. The dependent variables will be measured: pain intensity by means of Analogue Scale Visual, the function through the Constant-Murley test, the Movement Range with Goniometer and the Pressure Threshold Pain with a pressure gauge brand Stech.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years.
* Present clinical diagnosis of Subacromial Impingement Syndrome
* Threshold of pain in the Teres Major muscle pressure less than 2 Kg / cm2.
* Signature of informed consent.

Exclusion Criteria:

* Pre-shoulder surgery (<1 year).
* Inability to keep supine position.
* Contraindications for stretching: (collagen / tissue diseases connective: Ehlers-Danlos, Morquio, Grisel), scars in the healing process or pathological in the area like keloids, acute inflammatory process on the shoulder (<7 days), severe limitation of the range of movement towards flexion (<90º passive).
* Infiltrations (the last 3 months) or during treatment.
* Be pending litigation or legal claim.
* Cognitive problems or idiomatic barrier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2020-05-20 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 2 minutes needed for the explanation and the realization of the measure.
  It will be measured using an Analog Visual Scale. The scale to be used, always the same in each measurement.
Threshold Pressure Pain | 5 minutes needed for explain the technique and realise it.
  The patient will be placed in a chair with a table in front, where can support the elbow and forearm in shape comfortable. The physiotherapist takes a clamp without pushing the Teres Major muscle and will perform progressive pressure with the algometer until the patient refers pain sensation.
  The subjects who perceive pain with a threshold of pressure below 2kg / cm2 will be included in the study according to Andersen et al
Active Mobility | 10 minutes needed for explain the movements required and make de measurements.
  The measurement of active mobility (active flexion, active extension, active abduction, active external rotation, active internal rotation) will be done in standing position with the back supported in the framework of a door (to unify positions and allow us to carry out the extension) with a goniometer for flexion, extension, abduction and external rotation, and with a tape metric for internal rotation (measurement from the thumb to the spinous process of C7)
Function | 10 minutes needed for the realization of the test
  The assessment of the function will be performed through the constant Constant-Murley test.
  The Constant-Murley test abbreviated is a scale that measures the function of the shoulder on the basis of three components: pain, mobility and activities of daily life, resulting in a value maximum of 75 points, in the case that there is no limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma G Nin, Ms, Principal Investigator — Institut Català de la Salut
Locations (1):
- Centre de Rehabilitació en Atenció Primària (Institut Català de la Salut), Cornellà de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data can be shared once the study has finished and its subsequent publication with anyone who requires it formally in writing to the Main Investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual Participant Data will be available after its publication. Please contact the Main Investigator

REFERENCES:
- [Background] van der Heijden GJ. Shoulder disorders: a state-of-the-art review. Baillieres Best Pract Res Clin Rheumatol. 1999 Jun;13(2):287-309. doi: 10.1053/berh.1999.0021. PMID 10952865
- [Background] Page MJ, Green S, Mrocki MA, Surace SJ, Deitch J, McBain B, Lyttle N, Buchbinder R. Electrotherapy modalities for rotator cuff disease. Cochrane Database Syst Rev. 2016 Jun 10;2016(6):CD012225. doi: 10.1002/14651858.CD012225. PMID 27283591
- [Background] Yu H, Cote P, Shearer HM, Wong JJ, Sutton DA, Randhawa KA, Varatharajan S, Southerst D, Mior SA, Ameis A, Stupar M, Nordin M, van der Velde GM, Carroll L, Jacobs CL, Taylor-Vaisey AL, Abdulla S, Shergill Y. Effectiveness of passive physical modalities for shoulder pain: systematic review by the Ontario protocol for traffic injury management collaboration. Phys Ther. 2015 Mar;95(3):306-18. doi: 10.2522/ptj.20140361. Epub 2014 Nov 13. PMID 25394425
- [Background] van den Dolder PA, Roberts DL. A trial into the effectiveness of soft tissue massage in the treatment of shoulder pain. Aust J Physiother. 2003;49(3):183-8. doi: 10.1016/s0004-9514(14)60238-5. PMID 12952518
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738